CLINICAL TRIAL: NCT00204386
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Determine the Efficacy and Safety of Topiramate in the Treatment of Posttraumatic Stress Disorder
Brief Title: Safety & Efficacy Study Using Topiramate in Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPSS-205; IRB#10198
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study was to determine if Topiramate was safe and effective for use in civilian subjects with Posttraumatic Stress Disorder.

DETAILED DESCRIPTION:
Civilian PTSD is a widespread psychiatric condition and is commonly underestimated in terms of prevalence and morbidity, at least in the United States and probably world-wide. The magnitude of the public health impact of PTSD is highlighted by recent epidemiologic findings. Kessler, et al, estimated a 7.8% lifetime prevalence for PTSD in a representative national sample of 5877 persons aged 15-54. In part, this high prevalence is due to the high occurrence of trauma exposure over a lifetime. Common types of Civilian PTSD include serious physical attack or assault, rape, sexual assault, transportation accidents, exposure to death/homicide or serious injury, life-threatening accidents, threats of injury with fire, floods, weapons, natural disasters and civilian exposure to military attacks. Persons with PTSD are usually unaware that they have this disorder and because treatment professionals have been inadequately sensitized to high prevalence of this condition, the condition is markedly undiagnosed and thereby undertreated. The risk of PTSD is not restricted to the psychiatric population. In general, persons with PTSD seek help in general medical and not mental health settings. Individuals with PTSD are at increased risk of co-morbid psychiatric disorders including depression, alcohol and drug abuse, panic disorder, agoraphobia and personality disorders. It is associated with a substantially higher suicide risk, hospitalization rates, and increased utilization rates of non-psychiatric medical services as well as mental health services.

ELIGIBILITY:
Inclusion Criteria:

* PTSD as defined by DSM-IV for at least 6 months supported by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I);
* Subjects must have a minimum past week CAPS score of > than 50 at Visit 2;
* Subjects must be in general good health as confirmed by medical history, and physical examination;
* Subjects must be off prohibited medications for washout periods as outlined under Concomitant Therapy section;
* Subjects must have negative urine drug screen (phencyclidine, cocaine, amphetamines, tetrahydrocannabinol, and opiates) at visit 1;
* Subjects must either be postmenopausal for at least 1 year,have had a hysterectomy or tubal ligation, be otherwise incapable of pregnancy or have practiced one of the following methods of contraception for at least one month prior to enrollment: hormonal contraceptives, spermicide and barrier, intrauterine device, spousal/partner sterility or be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence.
* Subjects must be able to take oral medication, adhere to medication regiments and be willing to return for regular visits;
* After full explanation of the study, subjects must demonstrate their willingness to participate by signing an informed consent form.

Exclusion Criteria:

* Subjects who have a DSM-IV diagnosis of substance dependence or abuse (with the exception of nicotine or caffeine dependence) within the past 3 months;
* Subjects with current or past history of primary major depressive disorder or primary major anxiety disorder (i.e. panic disorder, obsessive-compulsive disorder, social phobia) as defined by DSM-IV;
* Subjects with current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder;
* Subjects with diagnosis of current organic mental disorder, factitious disorder or malingering
* Subjects with diagnosis of bulimia or anorexia nervosa;
* Subjects who are currently enrolled in cognitive-behavioral therapy;
* Subjects with current disability compensation or claim pending for persisting functional impairment related to PTSD;
* Subjects with prior non-response to topiramate for the treatment of PTSD following an adequate trial.
* Subjects who have previously been treated with topiramate and discontinued treatment due to an adverse event or subjects with a known hypersensitivity to topiramate;
* Subjects with clinically unstable disease: cardiovascular, renal, gastrointestinal, pulmonary, metabolic, endocrine or other systemic disease that could interfere with their participation in the study;
* Subjects with history of nephrolithiasis;
* Subjects with SGOT and/or SGPT levels greater than 2 times the upper limit of normal range at screening;
* Subjects taking antipsychotics within 3 months of the screening visit;
* Subjects with progressive or degenerative neurologic disorders (e.g. multiple sclerosis);
* Subjects with active liver disease;
* Subjects with estimated creatinine clearance < 60 mL/min;
* Subjects with known clinically significant medical conditions, including but not limited to: symptomatic coronary artery or peripheral vascular disease, malignancy within the past 5 years, except basal cell carcinoma; any condition compromising the function of those body systems that could result in altered absorption, excess accumulation or impaired metabolism or excretion of topiramate; subjects with history of attempted suicide/homicide in the past 12 months or suicidal/homicidal tendencies or judged clinically to be at serious suicidal/homicidal risk;
* Subjects who are pregnant or lactating;
* Subjects who have not observed the designated washout periods for any of the prohibited medications outline in this protocol;
* Subjects who in the opinion of the investigator should not be enrolled in the study because of the Precautions, Warnings, or Contraindications of the topiramate package insert.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2002-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Total CAPS Scale Score change from baseline/visit 2. CAPS administered at 5,7 and 9 | 12 weeks

SECONDARY OUTCOMES:
CGI Scale at visit 2 through 9; HARS at visit 2,4,5,7 and 9; HAM-D at visit 2,4,5,7 and 9; DTS at visits 2,4,5,7 and 9; TOP 8 at visits 2, 4-9; SDS visits 2-9; SVS visits 2-9 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Phebe M Tucker, MD, Principal Investigator — Professor
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States